CLINICAL TRIAL: NCT05481073
Title: Pilot Feasibility Study of Using UV Sensor in Patients With Actinic Keratosis
Brief Title: UV Sensor in Patients With Actinic Keratosis
Status: Completed | Type: Observational
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: Usability UV sensor study
Record Dates: First submitted 2022-06-22; First posted 2022-08-01 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Keratosis, Actinic
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: UV sensor — Use of UV sensor to be informed about the sun exposure daily through a mobile application

SUMMARY:
To validate the use of Ultraviolet (UV) radiation sensor in patients with actinic keratosis, to identify barriers to its use in prospective longitudinal studies.

DETAILED DESCRIPTION:
To prevent both acute and chronic damage from exposure to UV A and UV B radiation. Personal UV exposure can be assessed by portable sensors. Having an accurate awareness of one's own behavior (assessed by the accuracy of the UV sensor), can motivate and engage with skin protection.

ELIGIBILITY:
Inclusion Criteria:

>=65 years presenting actinic keratosis on scalp and/or face

Exclusion Criteria:

Patients who, due to health problems or lifestyle habits, do not expose themselves regularly to UV radiation (outdoor) for at least one hour a day.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Non-hospitalized patients routinely seen in dermatology outpatient clinics who meet the inclusion criteria will be offered the possibility of participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
QOL UV sensor | Up to week 4
  Questionnaire will be carried out to qualitatively evaluate different aspects of the usability of the UV device, Minimum Value 0; Maximun Value 20, where higher value is the better.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Unit (Hospital Clinic), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No